CLINICAL TRIAL: NCT06222879
Title: A Multi-center, Open-label Phase Ib/II Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of HRS-8080 or SHR-A2009 Combined With Anti-tumor Therapy in Patients With Unresectable or Metastatic Breast Cancer
Brief Title: Study of HRS-8080 or SHR-A2009 Combined With Anti-tumor Therapy in Patients With Unresectable or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8080-202
Record Dates: First submitted 2023-12-04; First posted 2024-01-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Three parallel arms
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A (Experimental)
  Interventions: Drug: HRS-8080; SHR-A1811
- Part B (Experimental)
  Interventions: Drug: HRS-8080; SHR-A2009
- Part C (Experimental)
  Interventions: Drug: SHR-A2009; SHR-1316

INTERVENTIONS:
Drug: HRS-8080; SHR-A1811 — Participants will receive HRS-8080 and SHR-A1811
  Arms: Part A
Drug: HRS-8080; SHR-A2009 — Participants will receive HRS-8080 and SHR-A2009
  Arms: Part B
Drug: SHR-A2009; SHR-1316 — Participants will receive SHR-A2009 and SHR-1316
  Arms: Part C

SUMMARY:
This study is designed to determine if treatments with the combination of HRS-8080 and SHR-A1811, the combination of HRS-8080 and SHR-A2009, the combination of SHR-A2009 and SHR-1316 are safe, tolerable, and has anti-cancer activity in patients with unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females aged 18-75 years old (both ends inclusive);
2. ECOG performance status (PS) 0-1 points;
3. Patients with metastatic or locally advanced breast cancer confirmed by histology（ER positive, HER2 positive/negative，or triple negative breast cancer）.
4. Tumor tissue samples must be provided for detection of tumor markers;
5. Menopausal state;
6. Disease progression confirmed by imaging during or after the last systemic treatment before enrollment;
7. There must be at least one measurable extracranial lesion that complies with RECIST v1.1;
8. Expected survival >3 months;
9. Good functional level of the organs ;
10. Female subjects with childbearing potential must agree to use highly effective contraceptive measures during the study treatment period and within 7 months after the end of the study treatment period; female subjects with childbearing potential must agree to use serum serum within 7 days before study enrollment. The HCG test must be negative and the patient must be non-lactating;
11. Voluntarily participate in this clinical trial, be willing and able to comply with clinical visits and research-related procedures, understand the research procedures and have signed informed consent.

Exclusion Criteria:

1. Patients with active (without medical control or clinical symptoms) brain metastasis;
2. Have the following lung diseases or history;
3. History of clinically severe cardiovascular disease;
4. Those who have received immunosuppressants or systemic hormone therapy for immunosuppression within 2 weeks before the first dose (dose >10 mg/d prednisone or other corticosteroids at equivalent physiological doses), excluding nasal spray or inhaled hormones;
5. The damage caused by the subject receiving other treatments has not recovered (severity level NCI-CTCAE V5.0 classification ≤1, excluding hair loss and other adverse events judged to be tolerable by the researcher);
6. There are serious infections within 4 weeks before the first medication;
7. Untreated active hepatitis;
8. The subject has suffered from other malignant tumors in the past 5 years or currently, excluding cured cervical carcinoma in situ, cutaneous basal cell carcinoma and squamous cell carcinoma;
9. Presence of active autoimmune disease;
10. Have a history of immunodeficiency, including acquired (HIV infection), congenital immunodeficiency diseases, or a history of organ transplantation (including allogeneic bone marrow transplantation);
11. The subject is in the acute infection stage or active tuberculosis and requires drug treatment;
12. Known to be allergic to the components of HRS-8080, SHR-A1811 and its components, SHR-A2009 and its components, and Adebrelimab; have a history of severe allergic reactions to other monoclonal antibodies;
13. Patients who have other serious physical or mental illnesses or laboratory test abnormalities that may increase the risk of participating in the study or interfere with the results of the study, and who the researcher believes are not suitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity（DLT） | up to 1 cycle (21 days)
  Phase 1
Maximum Tolerable Dose（MTD） | up to 1 cycle (21 days)
  Phase 1
Recommended Phase 2 Dose（RP2D） | up to 1 cycle (21 days)
  Phase 1
Safety endpoints: the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) (rated based on CTCAE V5.0) | up to 12 months
  Phase 1
Efficacy endpoint: objective response rate (ORR) | up to 12 months
  Phase 2

SECONDARY OUTCOMES:
level of SHR-A1811 ADA and Nab | up to 12 months
  Phase 1
level of SHR-A2009 ADA and Nab | up to 12 months
  Phase 1
level of adebrelimab ADA and Nab | up to 12 months
  Phase 1
Objective response rate (ORR) | up to 12 months
  Phase 1
Best overall response (BOR) | up to 12 months
  Phase 1
Duration of response (DoR) | up to 12 months
  Phase 1
Disease control rate (DCR) | up to 12 months
  Phase 1
Clinical benefit rate (CBR) | up to 12 months
  Phase 1
Progression-free survival (PFS) | up to 12 months
  Phase 1
Safety endpoints: incidence and severity of AEs and SAEs (rated based on CTCAE V5.0) | up to 12 months
  Phase 2
level of SHR-A1811 ADA and Nab | up to 12 months
  Phase 2
level of SHR-A2009 ADA and Nab | up to 12 months
  Phase 2
level of adebrelimab ADA and Nab | up to 12 months
  Phase 2
Best overall response (BOR) | up to 12 months
  Phase 2
Duration of response (DoR) | up to 12 months
  Phase 2
Disease control rate (DCR) | up to 12 months
  Phase 2
Clinical benefit rate (CBR) | up to 12 months
  Phase 2
Progression-free survival (PFS) | up to 12 months
  Phase 2

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided